CLINICAL TRIAL: NCT03470558
Title: Role of Dietary Habits in Efficacy of Bariatric Surgery - Study A
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2017P002526A; R01HL140574 (NIH)
Record Dates: First submitted 2018-03-12; First posted 2018-03-20 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Bariatric Surgery; Sleeve Gastrectomy; Obesity
Keywords: Diet; Dietary Habits; Weight changes
MeSH Terms: conditions — Obesity; Feeding Behavior; Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Optional tissue collection during bariatric surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleeve gastrectomy patients: Patients electing to undergo sleeve gastrectomy will monitor their dietary habits.
  Interventions: Other: Dietary habits

INTERVENTIONS:
Other: Dietary habits — Sleeve gastrectomy patients will be asked to monitor dietary habits before surgery and at 2, 6, and 12 months after surgery.

SUMMARY:
The purpose of the study is to evaluate how dietary habits in the post-surgical year impact outcomes of bariatric surgery.

DETAILED DESCRIPTION:
The obesity epidemic is a major public health concern with a significant economic burden in the USA. Bariatric surgery is the most effective and durable weight loss treatment, with long-term cardiometabolic health benefits. Among different types of bariatric procedures, sleeve gastrectomy (SG) has become the most commonly performed in USA. While SG is expected to result in a 50-60% excess weight loss, inter-individual differences in weight loss are large and approximately 25% of patients can be considered poor weight-loss responders who either do not lose a substantial amount of weight or regain the lost weight afterwards. The mechanisms underlying this clinical variation remain unknown and interventions to improve on these outcomes critically lacking. Of interest, altered daily dietary habits are experienced by a substantial proportion of bariatric surgery candidates, raising the question whether such alterations may contribute to inter-individual differences in weight loss success. Therefore, the purpose of this study is to evaluate how dietary habits in the post-surgical year impact outcomes of bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery (sleeve gastrectomy) patients

Exclusion Criteria:

* Prior bariatric surgical procedures

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients electing to undergo sleeve gastrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change in BMI at 1-year post-surgical | Baseline and one year
  Body mass index at one year after surgery compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frank Scheer, PhD, Principal Investigator — Brigham and Women's Hospital; Ali Tavakkoli, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No